CLINICAL TRIAL: NCT00577083
Title: Cap-fitted Colonoscopy: a Randomized, Tandem Colonoscopy Study of Adenoma Miss Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 0501-30
Record Dates: First submitted 2007-12-11; First posted 2007-12-19 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2017-03

CONDITIONS: Polyps
Keywords: miss rates
MeSH Terms: conditions — Polyps | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Initial cap-fitted (Experimental): Initial cap-fitted colonoscopy for the first insertion
  Interventions: Device: Cap-fitted colonoscopy
- Initial regular (Active Comparator): Initial regular no cap on the end of the colonoscope for the first insertion
  Interventions: Device: Cap-fitted colonoscopy

INTERVENTIONS:
Device: Cap-fitted colonoscopy — Subjects will be randomized to either initial cap-fitted colonoscopy or regular colonoscopy. Patients in the initial regular arm, will undergo cap-fitted colonoscopy for their second, tandem examination. Patients in the initial cap-fitted arm, will under undergo regular colonoscopy (without the cap) for their second, tandem examination.
  Other Names: cap-assisted colonoscopy; colonoscopy with detachable hood

SUMMARY:
This is a test in which a thin, black, flexible tube with a lighting system on the end is passed through the anus, into the rectum, in order to examine the large bowel or intestine, also called the colon. Colonoscopy is a very good test for examining the colon for polyps (warty growths that can turn into cancer), but it is not perfect. In fact, about 30% of polyps that are under 5 mm (about 1/5 of an inch) in size are missed during colonoscopy because they are hiding behind folds and bends in the colon. This research study is being done to determine if performing colonoscopy with a cap on the tip of the colonoscope will reduce the miss rate for polyps. A cap is a clear plastic hood that fits on the tip of the colonoscope and sticks out about 1/3 of an inch. During colonoscopy, the cap can be pressed against a fold or ridge in order to flatten it, so that the lining on the other side can be more easily seen. This may reduce the miss rate for colon polyps.

DETAILED DESCRIPTION:
Patient will undergo tandem colonoscopy on the same day using propofol sedation. Patients will undergo one colonoscopy without the cap and a second colonoscopy with the cap on. We will endeavor to keep the total examination time equal between the groups and approximately six minutes. The order in which patients receive the two colonoscopies (i.e. cap or without cap first) will be randomized. Any polyps detected during the first colonoscopy will be removed during that procedure. During the withdrawal phase, the time for examination will be measured with a stopwatch, and the stopwatch will be stopped at any time a polyp is located and restarted when the polyp has been removed and retrieved. The stopwatch will also be stopped for suctioning fluid or washing debris from the colon surface. Any polyp detected and removed during the first colonoscopy will be counted as the detection for that procedure. During the second colonoscopy, all polyps will also be removed when detected. Any polyp identified and removed during the second procedure will be counted as a miss for the first procedure. All polyps will be sent separately for pathologic evaluation. The time required to remove and retrieve polyps with and without the cap on will be measured using a stopwatch as a secondary end point. The primary end point will be the miss rate for colonoscopy with the cap and colonoscopy without the cap.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older, undergoing scheduled colonoscopy and able to give informed consent.

Exclusion Criteria:

* Previous surgical resection of the colon or rectum
* American Society of Anesthesiology class III or higher
* Inflammatory bowel disease
* Current use of anticoagulants.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K Rex, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Medical Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hewett DG, Rex DK. Cap-fitted colonoscopy: a randomized, tandem colonoscopy study of adenoma miss rates. Gastrointest Endosc. 2010 Oct;72(4):775-81. doi: 10.1016/j.gie.2010.04.030. Epub 2010 Jun 25. PMID 20579648

RESULTS

PARTICIPANT FLOW:
Groups:
- No Cap First, Then Cap-fitted: no cap on the end of the colonoscope for the first insertion
  Cap-fitted colonoscopy: Subjects will be randomized to either initial cap-fitted colonoscopy or regular colonoscopy. Patients in the initial regular arm, will undergo cap-fitted colonoscopy for their second, tandem examination. Patients in the initial cap-fitted arm, will under undergo regular colonoscopy (without the cap) for their second, tandem examination.
- Initial Cap-fitted First, Then No Cap: Initial cap-fitted colonoscopy for the first insertion
  Cap-fitted colonoscopy: Subjects will be randomized to either initial cap-fitted colonoscopy or regular colonoscopy. Patients in the initial regular arm, will undergo cap-fitted colonoscopy for their second, tandem examination. Patients in the initial cap-fitted arm, will under undergo regular colonoscopy (without the cap) for their second, tandem examination.
Period: First Intervention (14 Days)
Arm/Group | No Cap First, Then Cap-fitted | Initial Cap-fitted First, Then No Cap
Started | 48 | 52
Completed | 48 | 52
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | No Cap First, Then Cap-fitted | Initial Cap-fitted First, Then No Cap
Started | 48 | 52
Completed | 48 | 52
Not Completed | 0 | 0
Period: Second Intervention (14days)
Arm/Group | No Cap First, Then Cap-fitted | Initial Cap-fitted First, Then No Cap
Started | 48 | 52
Completed | 48 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No Cap First, Then Cap Fitted: no cap on the end of the colonoscope for the first insertion
  Cap-fitted colonoscopy: Subjects will be randomized to either initial cap-fitted colonoscopy or regular colonoscopy. Patients in the initial regular arm, will undergo cap-fitted colonoscopy for their second, tandem examination. Patients in the initial cap-fitted arm, will under undergo regular colonoscopy (without the cap) for their second, tandem examination.
- Initial Cap-fitted First Then No Cap: Initial cap-fitted colonoscopy for the first insertion
  Cap-fitted colonoscopy: Subjects will be randomized to either initial cap-fitted colonoscopy or regular colonoscopy. Patients in the initial regular arm, will undergo cap-fitted colonoscopy for their second, tandem examination. Patients in the initial cap-fitted arm, will under undergo regular colonoscopy (without the cap) for their second, tandem examination.
- Total: Total of all reporting groups
Arm/Group | No Cap First, Then Cap Fitted | Initial Cap-fitted First Then No Cap | Total
Number analyzed (Participants) | 48 | 52 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 52 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 29 | 28 | 57
Region of Enrollment [Number; unit: participants]
  United States | 48 | 52 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Adenomas
Description: Cap Fitted Colonoscopy (CFC) may significantly reduced miss rates for colorectal adenomas, specifically for small adenomas. This study is the first North American study of any design and the largest tandem study of CFC. CFC is a safe, simple, and inexpensive technology that could improve the reliability of colonoscopy in detecting colorectal neoplasia. Additional study of CFC in Western populations is warranted.
Time Frame: after the second colonoscopy is completed
Measure: Number; unit: First Colonoscopy number of adenomas
Groups:
- Initial Regular: no cap on the end of the colonoscope for the first insertion
  Cap-fitted colonoscopy: Subjects will be randomized to either initial cap-fitted colonoscopy or regular colonoscopy. Patients in the initial regular arm, will undergo cap-fitted colonoscopy for their second, tandem examination. Patients in the initial cap-fitted arm, will under undergo regular colonoscopy (without the cap) for their second, tandem examination.
Arm/Group | Initial Cap-fitted | Initial Regular
Number analyzed (Participants) | 52 | 48
First Colonoscopy number of adenomas
  Number of adenomas detected at first colonoscopy | 83 | 89
  Number of adenomas detected at second colonoscopy | 28 | 44

2. Secondary Outcome: Time for Examination Will be Measured With a Stopwatch, and the Stopwatch Will be Stopped at Any Time a Polyp is Located and Restarted When the Polyp Has Been Removed and Retrieved.
Description: During the second colonoscopy, all polyps will also be removed when detected. Any polyp identified and removed during the second procedure will be counted as a miss for the first procedure. All polyps will be sent separately for pathologic evaluation. The time required to remove and retrieve polyps with and without the cap on will be measured using a stopwatch as a secondary end point. The primary end point will be the miss rate for colonoscopy with the cap and colonoscopy without the cap.
Time Frame: after 2nd colonoscopy was completed in 24hrs
Population: Patients aged 50 years or older who were able to give informed consent and were scheduled for elective colonoscopy at IUH were eligible for enrollment. Exclusion criteria were American Society of Anesthesiologists class III or higher, previous surgical resection of the colon or rectum, inflammatory bowel disease, and current use of anticoagulants.
Measure: Mean (Standard Error); unit: Minutes
Groups:
- Insertion Inspection Times (Standard): Standard Colonscopy
- Insertion Inspection Times (Cap-Fitted); Inspection Times (Cap-Fitted); Total Procedure Time (Cap-Fitted): Cap-Fitted
- Inspection Times (Standard); Total Procedure Time (Standard): Standard
Arm/Group | Insertion Inspection Times (Standard) | Insertion Inspection Times (Cap-Fitted) | Inspection Times (Standard) | Inspection Times (Cap-Fitted) | Total Procedure Time (Cap-Fitted) | Total Procedure Time (Standard)
Number analyzed (Participants) | 48 | 52 | 48 | 52 | 52 | 48
Minutes | 3.1 (0.2) | 3.2 (0.2) | 7.0 (0.1) | 7.0 (0.1) | 18.1 (0.8) | 20.5 (1.2)

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed.
Arm/Group | Initial Regular | Initial Cap-fitted
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No